CLINICAL TRIAL: NCT06926699
Title: RehAbilitatioN Versus Early Medial PaTellofemoral LIGament Reconstruction in Patients With Acute First-Time PateLlar DIslocation: A Pilot RanDomized ControllEd Trial
Brief Title: MPFL Reconstruction Versus Rehabilitation
Acronym: ANTI-GLIDE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Arthroscopy Association of North America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANTI-GLIDE; $25000 (Other Grant/Funding Number: Arthroscopy Association of North America)
Record Dates: First submitted 2025-04-11; First posted 2025-04-15 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Patellar (or Kneecap) Instability and Mal-alignment; Patellar Dislocation
Keywords: MPFL; Medial Patellofemoral Ligament Reconstruction; Patellar dislocation
MeSH Terms: conditions — Patella Fracture; Patellar Dislocation | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medial Patellofemoral Ligament Reconstruction (Experimental): An initial evaluation with a diagnostic knee arthroscopy is done to ensure there are no loose bodies or osteochondral lesions missed on MRI that require removal or fixation. Graft harvest and preparation is done using either an autograft or allograft tendon as per a shared decision-making approach between the surgeon and patient. A 2cm longitudinal incision is made over the anteromedial aspect of the patella and dissection done between the second and third layers. Fixation (variable depending on surgeon preference) is performed over the proximal half of the patella. Another skin incision is then made over the medial femoral epicondyle with a guide pin passed through Schottle's point. The proximal femoral cortex is then drilled overtop of the guide pin to a diameter equal to the graft diameter with the remainder of the femoral tunnel drilled to 4.5mm.The graft ends are tied to the patellar fixation and shuttled through the second and third layers and fixed to the femur.
  Interventions: Procedure: Medial Patellofemoral Ligament Reconstruction
- Rehabilitation (Active Comparator): Patients will be initially placed in a patellar stabilizing brace and told to remain non weight-bearing for the first two weeks. Subjects will be permitted to perform gentle ROM exercises while in the knee brace with progressive weight-bearing as tolerated permitted at the 2-week mark. Formal physiotherapy commences at 2-weeks post-enrollment, with a goal of return to activities or sport at 6-months post-enrollment.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Procedure: Medial Patellofemoral Ligament Reconstruction — An initial evaluation with a diagnostic knee arthroscopy is done to ensure there are no loose bodies or osteochondral lesions missed on MRI that require removal or fixation. Graft harvest and preparation is done using either an autograft or allograft tendon as per a shared decision-making approach between the surgeon and patient. A 2cm longitudinal incision is made over the anteromedial aspect of the patella and dissection done between the second and third layers. Fixation (variable depending on surgeon preference) is performed over the proximal half of the patella. Another skin incision is then made over the medial femoral epicondyle with a guide pin passed through Schottle's point. The proximal femoral cortex is then drilled overtop of the guide pin to a diameter equal to the graft diameter with the remainder of the femoral tunnel drilled to 4.5mm.The graft ends are tied to the patellar fixation and shuttled through the second and third layers and fixed to the femur.
  Arms: Medial Patellofemoral Ligament Reconstruction
Other: Rehabilitation — Patients will be initially placed in a patellar stabilizing brace and told to remain non weight-bearing for the first two weeks. Subjects will be permitted to perform gentle ROM exercises while in the knee brace with progressive weight-bearing as tolerated permitted at the 2-week mark. Formal physiotherapy commences at 2-weeks post-enrollment, with a goal of return to activities or sport at 6-months post-enrollment.
  Arms: Rehabilitation

SUMMARY:
This study involves patients between the ages of 16 and 25 and have been diagnosed with a first-time traumatic patellar dislocation within the past 3 months. McMaster University and the investigators are receiving compensation from the Arthroscopy Association of North America to cover the costs of conducting the study.

Dislocations of the kneecap or patella is often treated without surgery, however up to 50% of patients will unfortunately experience recurrent instability of the patella. These episodes can cause damage to the bones and cartilage in the knee, which can result in long-term knee pain or weakness. Therefore, there is increasing interest to consider treating the knee with surgery right away in this population.

The purpose of this study is to determine the effect of medial patellofemoral ligament (MPFL) reconstruction compared to rest and physical rehabilitation on the rate of repeat patella dislocation, pain, and knee function for patients with their first patellar dislocation. The investigators will follow patients for at least one year after assigned treatment is started. Outcomes will be measured using surveys and checking medical records over the course of the study. The pilot will test this research study on a smaller scale before conducting a larger study. Patients will not be asked to attend additional visits outside of their typical follow-up schedule with their doctor.

There will be 30 patients recruited in total for this pilot study. Not all patients diagnosed with a patellar dislocation will be eligible to participate. Participation will be required at 6 regularly scheduled appointments that patients would need to attend to see the surgeon (even if they were not in the trial), including the screening visit, surgery date (if randomized to that treatment), 2-week, 6-week, 3-month, 6-month, and 12-month follow-up visits. Patients will be asked how they feel via various questionnaires and should take no longer than 15-20 minutes to complete the research forms at each visit.

If patients agree to participate in this study, treatment will be determined by a process called randomization. Randomization means that the treatment the patient receives will be decided by chance like flipping a coin. Patients will have a 1-in-2 chance of receiving one of the following treatments:

DETAILED DESCRIPTION:
Patellar dislocation is a common orthopedic injury, with an overall incidence of acute first-time dislocation ranging between 2.3 and 23.2 per 100 000 person years, occurring often secondary to a non-contact flexion-rotation injury. The medial patellofemoral ligament (MPFL) is an hourglass shaped structure that originates on the superomedial aspect of the patella, and inserts onto the medial femoral epicondyle. This ligament is essential, as it serves as a primary checkrein to lateral patellar translation between 0-30 degrees of knee flexion. Surgical intervention often aims to replace this ligament to recreate this checkrein, in the form of MPFL reconstruction. Traditionally, patients who have sustained first-time patellar dislocations have been treated nonoperatively, and surgical intervention has mostly been reserved for patients with recurrent dislocations. However, the evidence behind this decision-making process is limited.

Specifically, a recently published a systematic review and meta-analysis comparing early MPFL reconstruction with rehabilitation, finding a pooled recurrent dislocation rate of 7% (95%CI 2-17%) in the reconstruction group compared to 30% (95%CI 25-36%) in the rehabilitation group. Another meta-analysis reported inferior rates of recurrent dislocation with rehabilitation (30%, 95%CI 25-36%) compared to acute MPFL repair (7%, 95%CI 3-12%). These findings were again found in the pediatric population, as reported by another meta-analysis published by our group, finding a pooled recurrent dislocation rate of 25.1% in the surgical group, compared with 46.4% in the conservative management group. When stratifying results by type of surgical procedure performed, the MPFL reconstruction group had a recurrent dislocation rate of 3.1% compared to that of other procedures, such as MPFL repair, lateral release, or medial imbrication, with a recurrent dislocation rate of 39.4%.

There have only been two prospective studies comparing MPFL reconstruction with rehabilitation for first-time dislocation. Based on the minimal number of adverse events, these studies demonstrated safety of early surgical intervention in first-time patellar dislocations, in addition to lower rates of recurrent patellar instability. However, allocation into treatment groups was not randomized in one study while the other study had a small sample size of only 39 patients which may bias and limit the applicability of the results.

This is a pilot randomized controlled trial (RCT) that will determine in patients under 25 years old with acute first-time patellar dislocations, the effect of early medial patellofemoral ligament (MPFL) reconstruction vs rehabilitation on recurrent dislocation rates, anterior knee pain, patient reported functional outcomes and complication rates at 12 months. The rationale for this trial is based on 1) the burden of patellar instability in the general population, 2) the high risk of progression to recurrent instability, 3) serious long-term, deleterious effects to the knee with recurrent instability, 4) the lack of definitive evidence or guidelines on the optimal treatment strategy in patients with these injuries, 5) promising results seen with early MPFL reconstruction in previous smaller studies, 6) lack of well-powered, high-quality, RCTs assessing early MPFL reconstruction after an acute first-time patellar dislocation patients. This trial is important and novel because it will provide surgeons with high-quality level I evidence to guide treatment decisions in patients with acute first-time patellar dislocations.

ELIGIBILITY:
Inclusion Criteria:

1. Males and female patients under the age of 25 inclusive but greater than 10 years of age inclusive
2. Patients with first-time traumatic lateral patellar dislocation presenting within 6 months from time of injury
3. Lateral patellar dislocation confirmed by radiography, MRI demonstrating sequela of lateral patellar dislocation after injury to the knee, demonstration of patellar apprehension, J-sign or patellar glide grade 3 or greater on physical exam following injury to the knee
4. Patients who have the ability to speak, understand, and read English
5. Provision of informed consent or parental consent

Exclusion Criteria:

1. Previous dislocation episodes or instability of the affected patella
2. Previous surgeries involving the affected knee
3. History or clinical exam findings of generalized ligamentous laxity (defined as Beighton score of 4 or more points)
4. TT-TG distance >20mm as determined by MRI
5. Evidence of severe trochlear dysplasia on MRI as determined by Dejour classification type D dysplasia
6. Loose bodies or osteochondral fractures as confirmed on MRI
7. A neurovascular injury of the affected leg
8. Patients who will likely have problems, in the judgment of the investigator, with maintaining follow-up
9. Any other reason(s) the investigator feels is relevant for excluding the patient
10. Patients requiring concomitant arthrotomy for osteochondral fracture fixation (however microfracture and arthroscopic loose body removal for loose bodies found on arthroscopic assessment are not exclusion criteria)

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrent dislocation and instability | 12 months post- start of intervention
  1. The rate of recurrent patellar dislocation at 12 months
  2. The rate of recurrent subjective instability at 12 months
  3. The rate of recurrent instability requiring surgical management at 12 months

SECONDARY OUTCOMES:
Visual Analogue Score (VAS) | 12 months post- start of intervention
  The VAS is one of the most commonly used pain rating scores in both research and clinical practice, it is an easy-to-use, validated, one-dimensional scale from 0-10
Kujala Anterior Knee Pain Scale | 12 months post- start of intervention
  The Kujala Anterior Knee Pain scale is a 13-item screening instrument used to assess patellofemoral pain in adolescents and young adults, with a variable ordinal response format. Total scores range from 0-100.
Banff Patellofemoral Instability Index 2.0 (BPII2.0) | 12 months post- start of intervention
  The Banff Patellofemoral Instability Index 2.0 (BPII 2.0) Score is a metric of quality of life with multiple domains and subdomains having participants rate items from 0-100
Tegner Activity Scale | 12 months post- start of intervention
  The Tegner activity scale is a numerical scale with each value (0-10) representing specific activities An individual participating in competitive sports has an activity level of 10. An individual participating in recreational sports has an activity level of 6. An individual on sick leave or disability pension due to knee problems has an activity of 0
Adverse Events | 12 months post- start of intervention
  Occurrence of adverse events such as patellar fracture, patellar cartilage lesion or other events (other than recurrent patellar dislocations), obtaining a subsequent MRI to evaluate for pathology, and secondary chondral injury not present on an initial MRI if recurrent MRI is performed
Recurrent Instability of the Patella score | 12 months post- start of intervention
  Will also aim to validate the Recurrent Instability of the Patella score, this will help determine which patients may benefit from surgical intervention for first-time dislocation by classifying their risk of recurrent dislocation as either low, intermediate, or high based on preoperative factors.
  The Recurrent Instability of the Patella score consists of four factors: age <25 years (worth 2 points), skeletal immaturity (worth 1 point), Dejour A-D dysplasia (worth 1 point), and TT-TG/patellar length >= 0.5 (worth 1 point), for a maximum score of 5. Scores of 0-1 are deemed as low risk, 2-3 as intermediate risk, and 4-5 points as high risk.

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to avoid risks of compromising patient confidentiality.